CLINICAL TRIAL: NCT00004773
Title: Study of Cardiac and Paroxysmal Abnormalities in Rett Syndrome
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: Baylor College of Medicine (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Other Study IDs: 199/11798; BCM-H2465
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1997-01

CONDITIONS: Rett Syndrome
Keywords: Rett syndrome; neurologic and psychiatric disorders; rare disease
MeSH Terms: conditions — Rett Syndrome; Neurologic Manifestations; Mental Disorders; Rare Diseases

SUMMARY:
OBJECTIVES: I. Evaluate electrocardiographic parameters, including QT and PR intervals and QRS morphology/duration, across clinical stages in patients with Rett syndrome.

II. Characterize abnormalities of cardiac conduction and repolarization. III. Assess arrhythmias, heart rate variability, and autonomic nervous system function in these patients using 24-hour Holter monitoring.

IV. Record events believed to represent seizures with video, electroencephalogram (EEG), and polygraph monitoring in patients who have more than 1 clinical seizure every 5 days.

V. Characterize these events with respect to clinical manifestations, EEG correlates, and other physiologic data.

VI. Determine the frequency of seizures vs. events without electrographic correlates in these patients.

VII. Determine whether Rett syndrome patients have characteristic or unique types of seizures and/or an epileptic syndrome.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients receive an electrocardiogram at baseline and every 6 months for 3 years. Clinical stage II patients undergo 24-hour Holter monitoring on the same schedule; age-matched controls are tested once.

A group of patients with more than 1 seizure or possible seizure every 5 days undergo 5-day continuous electroencephalogram/polygraphic/video monitoring, with respiratory effort assessment, end tidal carbon dioxide and oxygen saturation levels, and a seizure log.

ELIGIBILITY:
* Classical Rett syndrome meeting Rett Syndrome Diagnostic Work Group criteria
* Age-matched girls without neurologic or cardiac problems entered as controls

Min Age: 0 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 95
Dates: Start 1995-08; Study Completion 1997-06

CONTACTS AND LOCATIONS:
Overall Officials: Daniel G. Glaze, Study Chair — Baylor College of Medicine

REFERENCES:
- [Background] Glaze DG. Commentary: the challenge of Rett syndrome. Neuropediatrics. 1995 Apr;26(2):78-80. doi: 10.1055/s-2007-979728. No abstract available. PMID 7566458
- [Background] Glaze DG, Schultz RJ. Rett Syndrome: Meeting the Challenge of This Gender-Specific Neurodevelopmental Disorder. Medscape Womens Health. 1997 Jan;2(1):3. PMID 9746669
- [Background] Sekul EA, Moak JP, Schultz RJ, Glaze DG, Dunn JK, Percy AK. Electrocardiographic findings in Rett syndrome: an explanation for sudden death? J Pediatr. 1994 Jul;125(1):80-2. doi: 10.1016/s0022-3476(94)70128-8. PMID 8021793